CLINICAL TRIAL: NCT06006533
Title: Investigation of the Effects of Fascia Relaxation Techniques Applied to Plantar Flexor Muscles on Proprioception, Balance and Flexibility.
Brief Title: Fascia Release Techniques Applied to Plantar Flexor Muscles and Acute Efficacy of Kinesio Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar61
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Balance; Distorted; Fascia; Anomaly
Keywords: proprioception; flexibility; balance
MeSH Terms: conditions — Congenital Abnormalities | interventions — Massage

STUDY DESIGN:
Intervention Model Description: kinesio taping and percussive massage techniques
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesio taping (Experimental): kinesio taping Technique: It is used to provide support to the joint range of motion and tissues. It has a wide range of uses for purposes such as correcting functional disorders, healing, protecting, reducing pain and inflammation. There are differences in cutting shapes according to the applied area and the target to be achieved.
  Interventions: Other: taping
- percussive massage (Experimental): Percussive Massage Technique: It is one of the instrument-assisted soft tissue mobilization techniques that emerged as a result of combining the effects of traditional massage and vibration therapy. With the mechanical oscillation effect that occurs in the Percussive Massage Technique, the muscle fiber is stimulated and an increase in reflex activity is observed.
  Interventions: Other: massage

INTERVENTIONS:
Other: taping — Kinesio taping will be applied in accordance with the fascia correction technique, including the plantar flexor muscles, and it will be requested to stay on the skin for 3 days.
  Arms: kinesio taping
Other: massage — Percussive Massage will be applied to the posterior part of the sural fascia, including the plantar flexor muscles, 3 times a week for 5 minutes.
  Arms: percussive massage

SUMMARY:
The aim of this study; The aim of this study is to examine the effects of kinesio taping technique and percussive massage technique applied to plantar flexor muscles on proprioception, balance and flexibility in healthy individuals.

DETAILED DESCRIPTION:
The sample of the study will consist of healthy individuals who have not had any discomfort or surgical operation related to the lower extremity in the last 6 months. The demographic information of the individuals who agreed to participate in the study will be recorded and their written consent will be obtained. Participants will be divided into 2 groups as kinesio taping and Percussive Massage groups by randomization method. The dominant lower extremities of both groups will be applied. The Percussive Massage group will be applied to the posterior part of the sural fascia for 5 minutes, 3 times a week, including the plantar flexor muscles. In the kinesio taping group, taping will be done in accordance with the fascia correction technique, including the plantar flexor muscles, and it will be requested to stay for 3 days. Both groups will be evaluated before and after the application. Joint position sense test will be used to evaluate proprioception. In the evaluation of balance, the one-leg standing test will be considered. In the evaluation of flexibility; The flexibility of the hamstring, gastrocnemius, and plantar fascia will be examined. The Straight Leg Lift Test will be performed to look at the flexibility of the hamstring muscle. Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being between the ages of 18 and 60

Exclusion Criteria:

* Injury or surgery involving the lower extremity in the last 6 months
* having had an operation
* Malignancy, aneurysm, fever, infection, fracture, osteoporosis, rheumatoid arthritis, diabetes,
* coagulation disorder etc. myofascial release techniques are contraindicated
* have ailments
* Having any disorder that will affect balance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Joint Position Sense Test | 1 weeks
  The joint to be evaluated is passively brought to a certain angle and it is waited for 10 seconds so that the person can learn the position of the joint. The person is asked to actively bring the evaluated extremity back to this angle with the eyes closed. When the person completes the movement, the error degrees between the predetermined angles are determined and averaged.
One Leg Standing Test | 1weeks
  Persons are positioned on one leg, with their hands on their waists, in front of a visually determined target. The foot to be tested is on the ground. The raised foot should not touch the leg on the ground. Time is kept from standing on one leg. The time taken until the foot held above touches the other leg or is lowered to the ground is recorded.
Evaluation of Gastrocnemius Elasticity | 1 weeks
  The person to be evaluated is positioned by extending his legs so that the heel is in contact with the wall, without bending the knees. The person is asked to pull the ankle towards himself without removing the heel from the wall. The distance between the person's thumb and the wall is measured and recorded.
Evaluation of Plantar Fascia Flexibility | 1 weeks
  The person to be evaluated is positioned by extending his legs so that the heel is in contact with the wall, without bending the knees. The person is asked to pull the fingers back without separating the heel and metatarsal heads from the wall. The distance between the person's thumb and the wall is measured and recorded.
Straight Leg Lift Test | 1 weeks
  The person to be evaluated lies in the supine position without bending their knees. The person is asked to raise the leg to be evaluated to the point where he or she will feel a stretching sensation in the back of the thigh, keeping the knee straight. It is recorded by measuring with a goniometer or digital inclinometer.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze MAMUR, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Umraniye, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leabeater AJ, Clarke AC, James L, Huynh M, Driller M. Under the Gun: Percussive Massage Therapy and Physical and Perceptual Recovery in Active Adults. J Athl Train. 2024 Mar 1;59(3):310-316. doi: 10.4085/1062-6050-0041.23. PMID 37248364
- [Background] Biz C, Nicoletti P, Tomasin M, Bragazzi NL, Di Rubbo G, Ruggieri P. Is Kinesio Taping Effective for Sport Performance and Ankle Function of Athletes with Chronic Ankle Instability (CAI)? A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2022 Apr 29;58(5):620. doi: 10.3390/medicina58050620. PMID 35630037
- [Background] Cain MS, Ban RJ, Chen YP, Geil MD, Goerger BM, Linens SW. Four-Week Ankle-Rehabilitation Programs in Adolescent Athletes With Chronic Ankle Instability. J Athl Train. 2020 Aug 1;55(8):801-810. doi: 10.4085/1062-6050-41-19. PMID 32577737
- [Background] Williams S, Whatman C, Hume PA, Sheerin K. Kinesio taping in treatment and prevention of sports injuries: a meta-analysis of the evidence for its effectiveness. Sports Med. 2012 Feb 1;42(2):153-64. doi: 10.2165/11594960-000000000-00000. PMID 22124445
- [Background] Helly KL, Bain KA, Gribble PA, Hoch MC. The Effect of Plantar Massage on Static Postural Control in Patients With Chronic Ankle Instability: A Critically Appraised Topic. J Sport Rehabil. 2020 Oct 7;30(3):507-511. doi: 10.1123/jsr.2020-0092. PMID 33027760